CLINICAL TRIAL: NCT05451407
Title: Phase Ib Clinical Trial to Evaluate the Efficacy and Safety of TQB2618 Injection Combined With Toripalimab Injection in Patients With Advanced Melanoma
Brief Title: Efficacy and Safety of TQB2618 Injection Combined With Toripalimab Injection in Patients With Advanced Melanoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2618-Ib-01
Record Dates: First submitted 2022-06-21; First posted 2022-07-11 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2022-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2618 injection combined with Toripalimab injection (Experimental): TQB2618 injection combined with Toripalimab injection，21 days as a treatment cycle.
  Interventions: Drug: TQB2618 injection; Drug: Toripalimab injection

INTERVENTIONS:
Drug: TQB2618 injection — Humanized IgG4 mab targeting TIM-3
Drug: Toripalimab injection — Monoclonal antibody against Programmed death factor receptor 1

SUMMARY:
This study is an open, single-center, multi-cohort phase Ib exploratory study, and 50 subjects are planned to be enrolled to observe the objective response rate of each subject. The safety evaluation of this study adopts common terminology criteria for adverse events version (CTCAE) 5.0 to evaluate the adverse events of drugs. Efficacy was evaluated using response evaluation criteria in solid tumors version (RECIST) 1.1 for immune-based therapeutics criteria.

ELIGIBILITY:
Inclusion Criteria:

* 1 Age: 18-75 years old;ECOG PS score: 0~1;The expected survival is over 3 months
* 2 Patients with advanced melanoma diagnosed histologically and/or cytologically
* 3 At least one measurable lesion was confirmed according to RECIST 1.1 criteria
* 4 Major organs are functioning normally
* 5 Female subjects of reproductive age should agree to use contraceptive methods (such as intrauterine devices, birth control pills, or condoms) during the study period and for 6 months after the end of the study;Negative serum pregnancy/urine pregnancy test within 7 days prior to study enrollment and must be non-lactating subjects;Male subjects should agree to use contraception during the study and for six months after the end of the study period

Exclusion Criteria:

* 1 Present or present with other malignant tumors within 3 years prior to first use
* 2 Unalleviated toxicity above CTCAE grade 1 due to any prior treatment
* 3 Major surgical treatment and significant traumatic injury were performed within 28 days prior to initial administration
* 4 A wound or fracture that has not healed for a long time
* 5 Those who have a history of psychotropic drug abuse and can't get rid of it or have mental disorders
* 6 Subject with any severe and/or uncontrolled disease
* 7 Prior chemotherapy within 3 weeks prior to initial drug use, and prior radiotherapy or other antineoplastic drugs within 2 weeks prior to initial drug use
* 8 Those who have participated in and used other antitumor clinical trials within 4 weeks prior to the first drug use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | Initial administration up to 21 days
  Certain adverse events related to the test drug occurred within 1 treatment cycle (21 days) of the subjects' first dose
phase II recommended dose | At the end of phase I, 1 subject received the first dose up to 21 days
  Optimal tolerated dose determined after the end of phase 1
objective response rate | Baseline up to 96weeks
  The proportion of subjects with complete response (CR) and partial response (PR) whose tumor volume reduced to a predetermined value and maintained the minimum time limit (at the time of the next imaging evaluation)

SECONDARY OUTCOMES:
Progression-Free Survival | disease progression before death,no more than 100 months
  The time between the onset of first medication and disease progression (PD) or death before PD
Disease Control Rate | Baseline up to 96 weeks
  The ratio of disease control cases (Partial Remission+Complete Response+Partial Remission ) to total cases was calculated
Overall Survival | No more than 100 months from the beginning of the first dose to death
  From the time of the patient's first treatment to the time of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China